CLINICAL TRIAL: NCT06956014
Title: Multicenter, Double-blind, Randomized, Placebo-controlled Trial to Evaluate the Efficacy and Safety of the Full-spectrum Cannabis Extract VER-01 in Patients With Chronic Low Back Pain
Brief Title: Efficacy and Safety of VER-01 in the Treatment of Patients With Chronic Low Back Pain
Acronym: EXPAND
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Vertanical GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VER-CLBP-003
Record Dates: First submitted 2025-04-24; First posted 2025-05-02 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Chronic Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- VER-01 corresponding to 22.5 mg THC (Experimental)
  Interventions: Drug: VER-01
- VER-01 corresponding to 32.5 mg THC (Experimental)
  Interventions: Drug: VER-01
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: VER-01 — Standardized soft extract from Cannabis sativa DKJ127 L., cannabis flos (Cannabis flower), corresponding to 19 mg Δ9-Tetrahydrocannabinol (THC) per ml drug product
  Arms: VER-01 corresponding to 22.5 mg THC; VER-01 corresponding to 32.5 mg THC
Other: Placebo — Comparator without active ingredient
  Arms: Placebo

SUMMARY:
The aim of the trial is to prove the efficacy and safety of VER-01 corresponding to 22.5 mg or 32.5 mg THC compared to placebo in patients with chronic low back pain (CLBP) for whom drug treatment is indicated and previous optimized treatments with non-opioid analgesics have not led to sufficient pain relief or were unsuitable due to contraindications or intolerance.

ELIGIBILITY:
Inclusion Criteria:

* Chronic (≥ 6 months) pain in the lower back (between the 12th thoracic vertebra and lower gluteal folds). CLBP patients without a clear specific somatic cause, for which targeted therapy can have a positive effect on the course of the disease.
* Patients with indicated opioid drug treatment where previous optimized treatments with non-opioid analgesics (including combinations) have not led to sufficient pain relief or were unsuitable due to contraindications or intolerance

Exclusion Criteria:

* Any painful comorbidity which could, in the opinion of the investigator, interfere with the low back pain intensity assessment during the trial participation
* Pregnant or breastfeeding female patients
* Known history of previous or current severe psychiatric disorder as per DSM-5 (e.g., schizophrenia, bipolar disorder, severe anxiety disorder, psychotic disorder, post-traumatic stress disorder), or currently taking antipsychotic medication.
* Cardiovascular event or clinically significant cardiac dysfunction (e.g., congestive heart failure, myocardial ischemia, arrhythmias, poorly controlled high blood pressure, congenital long QT syndrome) within 12 months prior to Visit 1 or a cardiac disorder that, in the opinion of the investigator, would put the patient at risk of a clinically significant arrhythmia or myocardial infarction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Efficacy based on pain reduction | From Baseline to Treatment Week 12
  The primary endpoint is the absolute change in mean CLBP intensity measured on an 11-point numerical rating scale (NRS) at Treatment Week 12 compared to Baseline (Study Week -1).

IPD SHARING:
Plan to Share IPD: No